CLINICAL TRIAL: NCT04391686
Title: Resting Energy Expenditure of the COronaVirus (COVID19) Patient in Reanimation Context
Acronym: RECOVERY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-04
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Obesity
Keywords: resting energy expenditure; artificial nutrition
MeSH Terms: conditions — COVID-19; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID intensive care unit
  Interventions: Diagnostic Test: indirect calorimetry
- intensive care unit
  Interventions: Diagnostic Test: indirect calorimetry
- obesity
  Interventions: Diagnostic Test: indirect calorimetry

INTERVENTIONS:
Diagnostic Test: indirect calorimetry — to determine and compare the resting energy expenditure of each group

SUMMARY:
Compare the resting energy expenditure of COVID-19 patients (obese or non-obese) in intensive care unit with mechanical ventilation to a control group of non-COVID-19 intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

For the Ambulatory Obese Control Group, the inclusion criteria are:

* Age ≥ 18 years;
* Patient followed in the nutrition service;
* Patient who benefited from an indirect calorimetry whatever the indication between 01/01/20 and 31/12/2020;
* BMI> 30.

For the COVID Group and the Resuscitation Control Group, the inclusion criteria are:

* Age ≥ 18 years;
* Patient having undergone a resuscitation stay
* Patient on mechanical ventilation (intubated or tracheotomized) during their stay in intensive care;
* Patient having benefited from an indirect calorimetry upon arrival in intensive care;

Only for the COVID Group:

* Patient hospitalized in intensive care for COVID 19 infection diagnosed by a positive PCR via nasopharyngeal sampling or endotracheal aspiration.
* Patient who has not yet carried out his post-resuscitation visit;

Only for the Resuscitation Control Group:

- Patient hospitalized in intensive care for an indication other than an infectious cause.

Exclusion Criteria:

Non-inclusion criteria for the Ambulatory Obese Control Group:

* Person deprived of liberty;
* Person subject to legal protection measures;
* Patient's opposition to participate in research.

The non-inclusion criteria for the COVID Group and the Resuscitation Control Group:

* For patients intubated during the resuscitation stay Fi02> 70% which does not allow a correct interpretation of the calorimetry;
* Pregnancy ;
* Person deprived of liberty;
* Person subject to legal protection measures;
* Opposition of the patient or the person of trust to participate in the research.

Only for the COVID Group:

* Contraindication to indirect calorimetry (claustrophobia for post-resuscitation patients where calorimetry is performed with a mask);
* Contraindication to bioimpedancemetry (electronic implants, limb amputation, weight <30kg or> 300kg);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to resuscitation under mechanical ventilation and who have benefited from a first indirect calorimetry measurement via COSMED Q NRG within 48 hours after their admission are identified by the physicians of the resuscitation department. If these patients meet all the inclusion criteria, they will be notified to the center's investigators so that the latter can take the necessary steps to inform the patient or the confidential person about the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
The resting energy expenditure (in Kcal / 24h) measured by indirect calorimetry during the stay in intensive care. | baseline and 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: Vincent FLORENT, MD, PhD, Principal Investigator — Centre Hospitalier Arras
Locations (1):
- Arras general hospital, Arras, France